CLINICAL TRIAL: NCT04342715
Title: A Multicentre Observational Study to Assess Immune Response Status in Patients Before and After Treatment for Visceral Leishmaniasis
Brief Title: A Study to Assess Immune Response Status in Patients Before and After Treatment for Visceral Leishmaniasis
Status: Active, not recruiting | Type: Observational
Sponsor: University of York (Other)
Collaborators: University of Gondar (Other); Kenya Medical Research Institute (Other); Makerere University (Other); University of Khartoum (Other); European Vaccine Initiative (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Principal Investigator, Paul Kaye, Professor of Immunology, University of York
Other Study IDs: ImmStat@Cure (PK202001); RIA2016V-1640 (Other Grant/Funding Number: EDCTP)
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Visceral Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — Antimony Sodium Gluconate; Paromomycin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3mm skin biopsies whole blood diagnostic residue tissue aspirates (bone marrow, spleen or lymph node according to local procedures)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients who have a diagnosis of visceral leishmaniasis and will be treated with SSG/PM
  Interventions: Drug: Sodium stibogluconate / paramomycin
- Control: Healthy volunteers

INTERVENTIONS:
Drug: Sodium stibogluconate / paramomycin — Treatment with Sodium stibogluconate / paramomycin
  Groups: Patients

SUMMARY:
ImmStat@Cure is a multicentre observational study designed to assess the immune status of patients before and after treatment for visceral leishmaniasis. Forty patients and 30 controls will be recruited per site. The follow-up period is 6 months from the end of treatment.

DETAILED DESCRIPTION:
ImmStat@Cure will be undertaken at 4 treatment centres for leishmaniasis in East Africa; the Institute for Endemic Diseases, University of Khartoum, Khartoum, Sudan, the University of Gondar, Gondar, Ethiopia, Amudat Hospital, Amudat, Uganda and the Kimalel and Chemolingot Health Centres, Baringo County, Kenya.

The primary objective of the study is to assess systemic and skin immune responses and parasite load in patients before, and at end of treatment for visceral leishmaniasis.

Secondary objectives are:

1. To identify systemic and local immune correlates of treatment outcome
2. To evaluate parasite genotype in relation to immune response characteristics
3. To compare immunological and parasitological data across each site and determine possible correlates of progression to PKDL

The outcomes include data on immune cell phenotypes and function in peripheral blood and tissue, as determined using standard methods in immunology (e.g. flow cytometry, transcriptomics and histopathology) and parasite quantitation (e.g. PCR, histopathology). There will be qualitative and quantitative analysis of data across patient cohorts and between patients and controls.

Forty patients diagnosed with VL from each site will be included in the study. Patients must be willing and able to adhere to the study procedures and to give written informed consent. All patients will have been clinically and parasitologically confirmed as having visceral leishmaniasis (VL) and will receive one round of sodium stibgluconate/paramomycin (SSG/PM) treatment as per normal clinical practice and regional guidelines. Thirty healthy endemic controls will also be studied from each country.

For patients, confirmation of VL will be made by visual identification of parasites in stained tissue smears according to recommended diagnostic practice (using bone marrow, spleen or lymph node aspirates as clinically indicated and as per local procedures). Parasites will be isolated from residual tissue aspirate and genotyped. Where tissue aspirate is not a recommended or currently performed diagnostic procedure, parasites will be isolated where possible from blood and diagnosis confirmed by PCR.

The study requires two additional blood draws, one taken before treatment and the second taken at the end of treatment.

The study also requires two 3mm skin biopsies (taken from the back of the neck/shoulder), one taken prior to the beginning of treatment and the second taken at the end of treatment. Biopsies will be taken under local anaesthesia. Patients refusing skin biopsies can still be recruited into the study.

For healthy controls, 23mL of blood will be taken on a single occasion, for diagnostic purposes and to provide blood for immunological analyses.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to 50 years on the day of diagnosis
* Have confirmed diagnosis of VL and be judged suitable for treatment using a standard regimen of SSG/PM
* Willing and able to give written informed consent
* For adolescents aged 12 to 17 years on the day of screening, written informed consent from a parent must be obtained in addition to assent from the patient
* Without any other significant health problems as determined by medical history, physical examination, results of screening tests and the clinical judgment of a medically qualified Clinical Investigator
* Negative for malaria on blood smear
* Judged, in the opinion of a medically qualified Clinical Investigator, to be able and likely to comply with all study requirements as set out in the protocol

Exclusion Criteria:

The patient may not enter the study if any of the following apply:

* Has HIV, HBV or HBC
* Has previously had any form of leishmaniasis
* Pregnancy or lactating mothers
* Any confirmed or suspected immunosuppressive or immunodeficient state, including; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months
* Tuberculosis, leprosy, or severe malnutrition (severe malnutrition in adults defined as a BMI <18.5, and in adolescents (12-17yrs) as a Z score cut-off value of <-2 SD)
* Any other significant disease, disorder or finding, which, in the opinion of a medically qualified Clinical Investigator, may influence the result of the study, or the volunteer's ability to participate in the study
* Unlikely to comply with the study protocol

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with a confirmed diagnosis of VL and judged suitable for standard treatment regimen of SSG/PM.Patients will be recruited by active case detection.
  Controls will be recruited using convenient sampling method.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2022-05-22 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Immune cell phenotypes present in peripheral blood and tissue | 36 months
  Identification of immune cell phenotypes present in peripheral blood and tissue before and after treatment for VL.
Parasite load in skin | 36 months
  Identification of parasite load in skin biopsies from patients with VL

SECONDARY OUTCOMES:
Parasite genotype | 36 months
  Evaluate parasite genotype in relation to immune response characteristics
Immunological and parasitological data across sites | 36 months
  To compare immunological and parasitological data across and between sites and determine possible correlates of progression to PKDL.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kaye, PhD, Study Director — University of York
Locations (1):
- KEMRI, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No